CLINICAL TRIAL: NCT04984902
Title: Reduction of BK Viremia in Kidney Transplant Patients Using the Seraph 100 Microbind® Affinity (Seraph 100) Blood Filter
Brief Title: Reduction of BK Viremia in Kidney Transplant Patients
Acronym: CP026
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ExThera Medical Europe BV (Industry)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP026
Record Dates: First submitted 2021-04-21; First posted 2021-08-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Kidney Diseases; Kidney Transplant Infection; Kidney Transplant; Complications
Keywords: BK Virus
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: The primary objective is to demonstrate the reduction of BK viremia by treating kidney transplant patients with the Seraph 100 Microbind® Affinity Blood Filter from ExThera Medical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): Treatment with Microbind® Affinity Blood Filter
  Interventions: Device: Extracorporal therapy
- Control (No Intervention): Antibiotics

INTERVENTIONS:
Device: Extracorporal therapy — Extracorporal therapy
  Arms: Treatment

SUMMARY:
Reduction of BK Viremia by treating kidney transplant patients.

DETAILED DESCRIPTION:
a clinical investigation plan (CIP) for the "Reduction of BK viremia in kidney transplant patients using the Seraph 100 Microbind® Affinity (Seraph 100) Blood Filter" clinical study, where BK is an abbreviation of the name of the first patient whom the virus was isolated from in 1971. This clinical study is intended to evaluate the reduction of BK viremia by treating kidney transplant patients with the Seraph 100 Microbind® Affinity Blood Filter from ExThera Medical. This clinical study is sponsored by ExThera Medical Corporation.

This clinical study will be conducted in accordance with this CIP. All parties involved in the conduct of the clinical study will be qualified by education, training, or experience to perform their tasks and this training will be documented appropriately.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant patients with a BK-viraemia ≥ 10,000 IU/ml.
2. Be ≥ 18 years old and ≤ 90 years old
3. Existing hemodialysis access

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
3. Presence of comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
4. Have Child-Pugh Class C cirrhosis
5. Have platelet count <30.000/uL
6. Contraindications for heparin sodium for injection
7. Subjects demonstrating any contraindication for this treatment as described in the IFU
8. Patients without existing hemodialysis access

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in log 10 viral load | At day 0 and the following 3 treatments within five days after beginning with the first treatment.
  Time-weighted change from baseline in log10 viral load within five days after first treatment.

SECONDARY OUTCOMES:
Number of participants with leukopenia | At day 0 and the following 3 treatments within five days after beginning with the first treatment.
  Number of participants with leukopenia
Number of participants with increase in serum creatinine | At day 0 and the following 3 treatments within five days after beginning with the first treatment.
  Number of participants with increase in serum creatinine between the treatment days
Number of participants with inoperative hypotension | At 0 and the following 3 treatments within five days after beginning with the first treatment.
  Number of participants with inoperative hypotension per treatment period
Number of participants with decreasing haemoglobin measurements | At day 0 and the following 3 treatments within five days after beginning with the first treatment.
  Number of participants with decreasing haemoglobin measurements per treatment period

OTHER OUTCOMES:
N (%) of patients with treatment emergent adverse events | 2 months
  N (%) of patients with treatment emergent adverse events
Laboratory data | 2 months
  Laboratory data (Blood test, Hematology, chemistry and coagulation)
Vital signs score | 2 months
  Vital signs score
Physical examination score | 2 months
  Physical examination score

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Tyczynski, Dr., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR